CLINICAL TRIAL: NCT02006160
Title: Effects of Dalfampridine on Cognition in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ralph H.B. Benedict, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEU3270511E
Record Dates: First submitted 2012-06-06; First posted 2013-12-10 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Active Comparator): dalfampridine
  Interventions: Drug: dalfampridine
- control (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dalfampridine — 10 mg bid
  Other Names: Ampyra
  Arms: treatment
Drug: placebo — 10 mg bid
  Arms: control

SUMMARY:
Cognitive impairment is common in multiple sclerosis (MS) and has devastating impact on functional activities. There is great demand for medications that will enhance cognitive capacity in MS patients. To date, there is no evidence for improvement in cognition following treatment with aminopyridines, but the few studies on the topic included neuropsychological (NP) tests as secondary or tertiary outcomes, and were methodologically flawed. Dalfampridine may enhance cognition by direct pharmacological mechanisms, and should have effects on motor outcomes as in prior studies. By combining cognition and motor outcomes in the proposed study, the investigators will evaluate if the same patients with positive effects show beneficial responses on motor outcomes including physical activity and if such motor outcomes mediate and/or moderate cognitive improvements with dalfampridine

DETAILED DESCRIPTION:
3a. Patient Sample and Recruitment

Subjects will be consecutively selected from the Western New York (NY) region where the Baird MS Center and the Jacobs Neurological Institute are located. Patients will be interviewed and their records reviewed to assess for inclusion/exclusion. Patients will then be approached in the clinic or contacted by telephone and invited to participate in this clinical trial. The attached flier will also be used to directly advertise the study to patients. Patients who initiate contact with the researcher will be interviewed to assess eligibility.

Inclusion Criteria. Patients will be eligible for the study if they fulfill all the inclusion criteria specified below

1. Males/Females who are ≥ 18 years old and < 65 years old and are capable of understanding and complying with the protocol, including speaking and writing fluent English and having at least a 9th grade education.
2. Have a diagnosis of MS, as per revised McDonald's Criteria.
3. Have not received steroids in last thirty (30) days or a relapse in the last ninety (90) days, and whose MS is considered stable.
4. Impression of cognitive impairment as indicated by one of the following: (a) positive NP testing following diagnosis of MS as determined by board certified neuropsychologist or with z scores <-1.5 below expectation in at least one cognitive domain, or (b) informant Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) >28.
5. An Expanded Disability Status Scale (EDSS) of ≤ 6.5.
6. Have given written informed consent prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care.
7. Are capable of performing the requirements of a NP test battery including at least 20/70 near visual acuity by near vision chart, with correction allowed.
8. If female, must neither be pregnant nor breast-feeding and must either (a) be > 12 months post-menopausal or surgically sterilized, or (b) agree to use an acceptable method of birth control for the duration of the study. Abstinence will not be considered an acceptable method of birth control.

Exclusion Criteria. Patients will be excluded from the study if they meet any one or more of the exclusion criteria specified below:

1. Have cognitive deficits caused by concomitant medication usage or other significant neurological/psychological disease e.g. Alzheimer's disease, Parkinson's disease, stroke, transient ischemic attack, Vascular Dementia, Huntington's disease, traumatic brain injury or chronic central nervous system (CNS) infection
2. Have evidence of other medical cause(s) of cognitive impairment
3. Evidence of major mental illness predating the onset of MS
4. Have evidence of major depression as determined by a positive Beck Depression Index-Fast Screen (BDIFS) and clinician interview
5. Have report of uncontrolled or labile hypertension, tachycardia, cardiovascular or cerebrovascular disease
6. History of seizure disorder.
7. Optic neuritis within 6 months of enrollment.
8. Trigeminal neuralgia.
9. Prior exposure to aminopyridines.

Additional Exclusion Criteria for optional speech module. Patients will not be eligible for enrollment in the optional speech module is they meet one or more of the exclusion criteria below:

1. Have any language/dialect other than Standard American English as their first language.
2. Make use of a mechanical hearing aid.

3b. Outcome Measures

Cognition Endpoints. Psychometric testing will incorporate gold standard tests from validated test batteries by Benedict et al and Rao et al [7-9, 47-49]. The test order is described below:

Table 2. Cognitive Battery Test Domain Time in min California Verbal Learning Test 2 (CVLT2) Learning Trials Auditory/Verbal Memory 15 Brief Visuospatial Memory Test Revised (BVMTR) Learning Trials Visual/Spatial Memory 05 Paced Auditory Serial Addition Test (PASAT) 3 sec Auditory Processing Speed 05 Symbol Digit Modalities Test (SDMT) Visual Processing speed 05 Delis Kaplan Executive Function System (DKEFS) Sorting Test Executive Function 12 California Verbal Learning Test 2 (CVLT2) Delayed Recall Auditory/Verbal Memory 05 Brief Visuospatial Memory Test Revised (BVMTR) Delayed Recall Visual/Spatial Memory 03 Total Time 50 min

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if they fulfill all the inclusion criteria specified below:

1. Males/Females who are ≥ 18 years old and < 65 years old and are capable of understanding and complying with the protocol, including speaking and writing fluent English and having at least a 9th grade education.
2. Have a diagnosis of MS, as per revised McDonald's Criteria.
3. Have not received steroids in last thirty (30) days or a relapse in the last ninety (90) days, and whose MS is considered stable.
4. Impression of cognitive impairment as indicated by one of the following: (a) positive NP testing following diagnosis of MS as determined by board certified neuropsychologist or with z scores <-1.5 below expectation in at least one cognitive domain, or (b) informant MSNQ >28.
5. An Expanded Disability Status Scale (EDSS) of ≤ 6.5.
6. Have given written informed consent prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care.
7. Are capable of performing the requirements of a NP test battery including at least 20/70 near visual acuity by near vision chart, with correction allowed.
8. If female, must neither be pregnant nor breast-feeding and must either (a) be > 12 months post-menopausal or surgically sterilized, or (b) agree to use an acceptable method of birth control for the duration of the study. Abstinence will not be considered an acceptable method of birth control.

Exclusion Criteria:

1. Have cognitive deficits caused by concomitant medication usage or other significant neurological/psychological disease e.g. Alzheimer's disease, Parkinson's disease, stroke, transient ischemic attack, Vascular Dementia, Huntington's disease, traumatic brain injury or chronic CNS infection
2. Have evidence of other medical cause(s) of cognitive impairment
3. Evidence of major mental illness predating the onset of MS
4. Have evidence of major depression as determined by a positive BDIFS and clinician interview
5. Have report of uncontrolled or labile hypertension, tachycardia, cardiovascular or cerebrovascular disease
6. History of seizure disorder.
7. Optic neuritis within 6 months of enrollment.
8. Trigeminal neuralgia.
9. Prior exposure to aminopyridines within the last six months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Benedict, PhD, Principal Investigator — University at Buffalo; Bianca Weinstock-Guttman, MD, Principal Investigator — University at Buffalo
Locations (1):
- Buffalo General Hospital, Buffalo, New York, United States

REFERENCES:
- [Derived] Satchidanand N, Drake A, Smerbeck A, Hojnacki D, Kolb C, Patrick K, Weinstock-Guttman B, Motl R, Benedict RH. Dalfampridine benefits ambulation but not cognition in multiple sclerosis. Mult Scler. 2020 Jan;26(1):91-98. doi: 10.1177/1352458518815795. Epub 2018 Dec 19. PMID 30566030

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 45 | 16
Completed | 41 | 16
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 45 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 16 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.2) | 53 (7.5) | 49.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 10 | 48
  Male | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Symbol Digit Modalities Test
Description: The Symbol Digit Modalities Test is a measure of cognitive processing speed. The outcome is the total number of correct digit substitutions in 90 seconds, with a possible total range of 0-120. Higher values reflect a better score/outcome than lower scores.
Time Frame: Week 0, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 45 | 16
score on a scale
  Week 0 | 41.18 (10.67) | 35.06 (12.51)
  Week 12 | 45.05 (11.09) | 38.63 (10.82)

ADVERSE EVENTS:
Time Frame: From study Start to Study Completion (12 weeks per participant)
Description: The definitions do not differ from the clinicaltrials.gov definitions.
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/16
Other Adverse Events (participants affected / at risk) | 2/45 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=45) | Control (N=16)
Headache (General disorders) | 1 (1) | 0 (0) — Headache
Dizziness (General disorders) | 2 (2) | NA — Dizziness
Tremors (General disorders) | 1 (1) | NA — Tremors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No